CLINICAL TRIAL: NCT02287311
Title: ADMINISTRATION OF MOST CLOSELY MATCHED THIRD PARTY RAPIDLY GENERATED LMP, BARF1 and EBNA1 SPECIFIC CYTOTOXIC T-LYMPHOCYTES TO PATIENTS WITH EBV-POSITIVE LYMPHOMA AND OTHER EBV-POSITIVE MALIGNANCIES
Brief Title: Most Closely Matched 3rd Party Rapidly Generated LMP, BARF1 And EBNA1 Specific CTL, EBV-Positive Lymphoma (MABEL)
Acronym: MABEL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Rayne Rouce, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-35253 MABEL; MABEL (Other: Baylor College of Medicine)
Record Dates: First submitted 2014-11-06; First posted 2014-11-10 (Estimated); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Hodgkin Disease; Non-Hodgkin Lymphoma; Severe Chronic Active Epstein Barr Virus; T/NK-lymphoproliferative Disease; Nasopharyngeal Carcinoma; Smooth Muscle Tumor
Keywords: EBV positive diseases; cytotoxic T lymphocytes
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Nasopharyngeal Carcinoma; Smooth Muscle Tumor | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A: MABEL CTLs (Experimental): Patients with 1st or subsequent relapse.
  Three different dosing schedules will be evaluated. Two to four patients will be evaluated on each dosing schedule. Each patient will receive 2 injections, 14 days apart.
  If the patient's level of circulating T cells is relatively high, s/he may require treatment with cyclophosphamide (Cytoxan) and Fludarabine before s/he receives MABEL CTLs.
  Interventions: Biological: MABEL CTLs; Drug: Cyclophosphamide; Drug: Fludarabine
- Group B: MABEL CTLs (Experimental): Patients with persistent active disease despite therapy.
  Three different dosing schedules will be evaluated. Two to four patients will be evaluated on each dosing schedule. Each patient will receive 2 injections, 14 days apart.
  If the patient's level of circulating T cells is relatively high, s/he may require treatment with cyclophosphamide (Cytoxan) and Fludarabine before s/he receives MABEL CTLs.
  Interventions: Biological: MABEL CTLs; Drug: Cyclophosphamide; Drug: Fludarabine
- Group C: MABEL CTLs (Experimental): Patients with active disease if immunosuppressive chemotherapy is contraindicated.
  Three different dosing schedules will be evaluated. Two to four patients will be evaluated on each dosing schedule. Each patient will receive 2 injections, 14 days apart.
  If the patient's level of circulating T cells is relatively high, s/he may require treatment with cyclophosphamide (Cytoxan) and Fludarabine before s/he receives MABEL CTLs.
  Interventions: Biological: MABEL CTLs; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: MABEL CTLs — Dose escalation:
  DL1:2x10^7 cells/m2+2x10^7 cells/m2
  DL2:2x10^7cells/m2+5x10^7 cells/m2
  DL3:5x10^7 cells/m2+1x10^8 cells/m2
  *Doses are based on total CD3+cells/m2
  Patients with active disease that have apparent clinical benefit at the 8 wk post 1st infusion (6 wks after 2nd infusion) or subsequent evaluations may receive up to 6 additional doses of CTLs at intervals at least 6 wks apart, each of which will consist of the same cell number as their second injection or below the original dose if there is not enough product available for the original dose. Patients may receive lymphodepleting chemotherapy (Cy/Flu) before additional infusions. Patients cannot receive additional doses until the initial safety profile is completed at 6 wks following the second infusion.
  Other Names: LMP, BARF-1 and EBNA1 specific cytotoxic T lymphocytes; MABEL Cytotoxic T cells
Drug: Cyclophosphamide — If the patient's level of circulating T cells is relatively high, s/he may require treatment with cyclophosphamide (Cytoxan) and Fludarabine before s/he receives MABEL CTLs.
  3 daily doses of cyclophosphamide (Cy: 500 mg/m2/day) together with fludarabine (Flu: 30 mg/m2) to induce lymphopenia, finishing at least 24 hours before CTL infusion.
  Other Names: Cytoxan
Drug: Fludarabine — If the patient's level of circulating T cells is relatively high, s/he may require treatment with cyclophosphamide and fludarabine before s/he receives MABEL CTLs.
  3 daily doses of cyclophosphamide (Cy: 500 mg/m2/day) together with fludarabine (Flu: 30 mg/m2) to induce lymphopenia, finishing at least 24 hours before CTL infusion.
  Other Names: Fludara

SUMMARY:
The subject has a type of cancer or lymph gland disease associated with a virus called Epstein Barr Virus (EBV), which has come back, is at risk of coming back, or has not gone away after standard treatments. This research study uses special immune system cells called LMP, BARF-1 and EBNA1- specific cytotoxic T lymphocytes (MABEL CTLs).

Some patients with Lymphoma (such as Hodgkin (HD) or non-Hodgkin Lymphoma (NHL)), T/NK-lymphoproliferative disease, or CAEBV, or solid tumors such as nasopharyngeal carcinoma (NPC), smooth muscle tumors, and leiomyosarcomas show signs of a virus called EBV before or at the time of their diagnosis. EBV causes mononucleosis or glandular fever ("mono" or the "kissing disease"). EBV is found in the cancer cells of up to half the patients with HD and NHL, suggesting that it may play a role in causing Lymphoma. The cancer cells (in lymphoma) and some immune system cells (in CAEBV) infected by EBV are able to hide from the body's immune system and escape destruction. EBV is also found in the majority of NPC and smooth muscle tumors, and some leiomyosarcomas. We want to see if special white blood cells (MABEL CTLs) that have been trained to kill EBV infected cells can survive in your blood and affect the tumor.

In previous studies, EBV CTLs were generated from the blood of the patient, which was often difficult if the patient had recently received chemotherapy. Also, it took up to 1-2 months to make the cells, which is not practical when a patient needs more urgent treatment. To address these issues, the MABEL CTLs were made in the lab in a simpler, faster, and safer way. The MABEL CTLs will still see LMP proteins but also two other EBV proteins called EBNA-1 and BARF. To ensure these cells are available for use in patients in urgent clinical need, we have generated MABEL CTLs from the blood of healthy donors and created a bank of these cells, which are frozen until ready for use. We have previously successfully used frozen T cells from healthy donors to treat EBV lymphoma and virus infections and we now have improved our production method to make it faster.

In this study, we want to find out if we can use banked MABEL CTLs to treat HD, NHL, T/NK-lymphoproliferative disease, CAEBV, NPC, smooth muscle tumors or leiomyosarcoma. We will search the bank to find a MABEL CTL line that is a partial match with the subject.

MABEL CTLs are investigational and not approved by the Food and Drug Administration.

DETAILED DESCRIPTION:
A healthy donor has given blood to make LMP/BARF1/EBNA-1 MABEL CTLs in the lab. We made the cells by first growing a special type of cells called activated T cells to stimulate the T cells. We then added specially produced mixtures of proteins that include the LMP, EBNA1 and BARF proteins. These were used to stimulate T cells. As the T cells grew, we added some of the healthy donor cells expressing these proteins to stimulate them. We also added a cell called K562 that has had new genes put inside it so it expresses proteins that stimulate the immune system to encourage the T cells to grow. K562 cells are cancer cells that have been treated with radiation so they cannot grow. This stimulation trained the MABEL CTLs to kill cells with EBV proteins on their surface. These cells were grown and frozen.

For the subject's treatment, the MABEL CTLs will be thawed and infused into the subject over 1-10 minutes. Initially, two doses of MABEL CTLs will be given two weeks apart. Subjects may be eligible to receive additional doses of the MABEL CTLs up to 6 times.

All of the treatments will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital.

Medical tests before treatment:

Before being treated, the subject will receive a series of standard medical tests:

Physical exam; Blood tests to measure blood cells, kidney and liver function; Tumor measurements by routine imaging studies: Computer Tomogram (CT), Magnetic Resonance Imaging (MRI), or Positron Emission Tomography (PET/CT); Pregnancy test for females who are able to have children.

Several studies suggest that the infused T cells need room to be able to proliferate and accomplish their functions and that this may not happen if there are too many other T cells in circulation. Because of that, if the patient's level of circulating T cells is relatively high, s/he may require treatment with cyclophosphamide (Cytoxan) and fludarabine before s/he receives MABEL CTLs.

Medical tests during and after treatment:

Blood tests to measure blood cells, kidney and liver function; Imaging study 8 weeks after the 1st CTL infusion. If the subject receives additional doses they will also have an imaging study at 1 to 3 months after their final dose.

Subjects will either be seen in the clinic or will be contacted by research staff yearly for 5 years.

ELIGIBILITY:
Inclusion Criteria:

SCREENING

1. Any patient regardless of age or sex, with diagnosis of either:

   * EBV positive Hodgkin's lymphoma
   * EBV Positive non-Hodgkin's Lymphoma (regardless of histologic subtype)
   * EBV (associated)-T/NK-lymphoproliferative disease
   * Severe Chronic Active EBV (CAEBV) -- CAEBV is defined as patients with high EBV viral load in plasma or PBMC (>4000 genomes per ug PBMC DNA) and/or biopsy tissue positive for EBV
   * Other EBV positive malignancies (e.g. nasopharyngeal carcinoma, smooth muscle tumors, etc.)

   AND
   * in first or subsequent relapse (Group A)
   * with active disease persisting despite therapy (Group B)
   * with active disease if immunosuppressive chemotherapy is contraindicated e.g. patients who develop Hodgkin disease after solid organ transplantation or if the lymphoma is a second malignancy e.g. a Richter's transformation of CLL. (Group C)
2. EBV positive tumor
3. Weighs at least 12kg
4. Informed consent (and assent as applicable) obtained from patient/guardian.

TREATMENT

1. Any patient regardless of age or sex, with diagnosis of either:

   * EBV positive Hodgkin's lymphoma
   * EBV Positive non-Hodgkin's Lymphoma (regardless of histologic subtype)
   * EBV (associated)-T/NK-lymphoproliferative disease
   * Severe Chronic Active EBV (CAEBV) -- CAEBV is defined as patients with high EBV viral load in plasma or PBMC (>4000 genomes per ug PBMC DNA) and/or biopsy tissue positive for EBV
   * Other EBV positive malignancies (e.g. nasopharyngeal carcinoma, smooth muscle tumors, etc.)

   AND
   * in first or subsequent relapse (Group A)
   * with active disease persist despite therapy (Group B)
   * with active disease if immunosuppressive chemotherapy is contraindicated e.g. patients who develop Hodgkin disease after solid organ transplantation or if the lymphoma is a second malignancy e.g. a Richter's transformation of CLL. (Group C)
2. EBV positive tumor
3. Patients with life expectancy greater than or equal to 6 weeks
4. Patients with bilirubin less than or equal to 3x upper limit of normal
5. AST less than or equal to 5x upper limit of normal
6. Hemoglobin greater than or equal to 7.0 (may be a transfused value)
7. Patients with a creatinine less than or equal to 2x upper limit of normal for age
8. Pulse oximetry of > 90% on room air
9. Patients should have been off other investigational therapy for 30 days prior to infusion.
10. Patients with a Karnofsky/Lansky score of more than or equal to 50.
11. Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. The male partner should use a condom.
12. Informed consent (and assent as applicable) obtained from patient/guardian.

Exclusion Criteria:

TREATMENT

1. Pregnant or lactating
2. Severe intercurrent infection
3. Current use of systemic corticosteroids more than 0.5 mg/kg/day
4. Patients receiving ATG, Campath, or other immunosuppressive T cell monoclonal antibodies within 30 days.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-02; Primary Completion 2024-01-12 (Actual); Study Completion 2029-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rayne H Rouce, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 38 enrolled participants, 2 were screened but did not receive EBV Specific T cell (EST) infusions as they opted for alternate treatment while 36 participants received at least one EST infusion across three treatment groups (A, B and C), with each group having three dose levels. One of the treated participants who was not evaluable for DLT and response, and later re-enrolled was counted as 2 individual participants for the purpose of reporting.
Groups:
- Group A Cohort 1: Group A: Participants with 1st or subsequent relapse.
  Cohort 1: Participants were administrated EBV Specific T cells (ESTs), consisting of two infusions 2x10^7 cells/m2 and 2x10^7 cells/m2,14 days apart.
- Group A Cohort 2: Group A: Participants with 1st or subsequent relapse.
  Cohort 2: Participants were administrated EBV Specific T cells (ESTs), consisting of two infusions 2x10^7cells/m2 and 5x10^7 cells/m2,14 days apart.
- Group A Cohort 3: Group A: Participants with 1st or subsequent relapse.
  Cohort 3: Participants were administrated EBV Specific T cells (ESTs), consisting of two infusions 5x10^7 cells/m2 and 1x10^8 cells/m2
  ,14 days apart.
- Group B Cohort 1: Group B:Participants with persistent active disease despite therapy.
  Cohort 1: Participants were administrated EBV Specific T cells (ESTs), consisting of two infusions 2x10^7 cells/m2 and 2x10^7 cells/m2,14 days apart.
- Group B Cohort 2: Group B:Participants with persistent active disease despite therapy.
  Cohort 2: Participants were administrated EBV Specific T cells (ESTs), consisting of two infusions 2x10^7cells/m2 and 5x10^7 cells/m2,14 days apart.
- Group B Cohort 3: Group B:Participants with persistent active disease despite therapy.
  Cohort 3: Participants were administrated EBV Specific T cells (ESTs), consisting of two infusions 5x10^7 cells/m2 and 1x10^8 cells/m2
  ,14 days apart.
- Group C Cohort 1: Group C: Participants with active disease if immunosuppressive chemotherapy is contraindicated.
  Cohort 1: Participants were administrated EBV Specific T cells (ESTs), consisting of two infusions 2x10^7 cells/m2 and 2x10^7 cells/m2,14 days apart.
- Group C Cohort 2: Group C: Participants with active disease if immunosuppressive chemotherapy is contraindicated.
  Cohort 2: Participants were administrated EBV Specific T cells (ESTs), consisting of two infusions 2x10^7cells/m2 and 5x10^7 cells/m2,14 days apart.
- Group C Cohort 3: Group C: Participants with active disease if immunosuppressive chemotherapy is contraindicated.
  Cohort 3: Participants were administrated EBV Specific T cells (ESTs), consisting of two infusions 5x10^7 cells/m2 and 1x10^8 cells/m2
  ,14 days apart.
Period: Cohort 1: Dose Level 1
Arm/Group | Group A Cohort 1 | Group A Cohort 2 | Group A Cohort 3 | Group B Cohort 1 | Group B Cohort 2 | Group B Cohort 3 | Group C Cohort 1 | Group C Cohort 2 | Group C Cohort 3
Started | 3 | 0 | 0 | 5 | 0 | 0 | 2 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 5 | 0 | 0 | 2 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 2: Dose Level 2
Arm/Group | Group A Cohort 1 | Group A Cohort 2 | Group A Cohort 3 | Group B Cohort 1 | Group B Cohort 2 | Group B Cohort 3 | Group C Cohort 1 | Group C Cohort 2 | Group C Cohort 3
Started | 0 | 3 (Cohort 2 started after Cohort 1 completed.) | 0 | 0 | 3 (Cohort 2 started after Cohort 1 completed.) | 0 | 0 | 4 (Cohort 2 started after Cohort 1 completed.) | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not Completed | 0 | 3 | 0 | 0 | 3 | 0 | 0 | 2 | 0
Not completed — Death | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Refused follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 3: Dose Level 3
Arm/Group | Group A Cohort 1 | Group A Cohort 2 | Group A Cohort 3 | Group B Cohort 1 | Group B Cohort 2 | Group B Cohort 3 | Group C Cohort 1 | Group C Cohort 2 | Group C Cohort 3
Started | 0 | 0 | 6 (Cohort 3 started after Cohort 2 completed.) | 0 | 0 | 7 (Cohort 3 started after Cohort 2 completed.) | 0 | 0 | 3 (Cohort 3 started after Cohort 2 completed.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 6 | 0 | 0 | 7 | 0 | 0 | 3
Not completed — Death | 0 | 0 | 4 | 0 | 0 | 4 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — On long-term follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one EST infusion will be included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A Cohort 1 | Group A Cohort 2 | Group A Cohort 3 | Group B Cohort 1 | Group B Cohort 2 | Group B Cohort 3 | Group C Cohort 1 | Group C Cohort 2 | Group C Cohort 3 | Total
Number analyzed (Participants) | 3 | 3 | 6 | 5 | 3 | 7 | 2 | 4 | 3 | 36
Age, Continuous [Median (Full Range); unit: years] | 15.0 [14.0 to 80.0] | 18.0 [17.0 to 20.0] | 18.5 [11.0 to 42.0] | 54.0 [7.0 to 72.0] | 51.0 [36.0 to 51.0] | 41.0 [4.0 to 61.0] | 36.0 [16.0 to 56.0] | 9.5 [7.0 to 34.0] | 37.0 [7.0 to 77.0] | 19.5 [4.0 to 80.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 11
  Male | 0 | 3 | 5 | 4 | 2 | 6 | 1 | 3 | 1 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 5
  Not Hispanic or Latino | 3 | 2 | 5 | 5 | 3 | 6 | 2 | 2 | 2 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 6
  White | 2 | 3 | 2 | 4 | 3 | 4 | 1 | 3 | 3 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Dose-limiting Toxicity (DLT)
Description: To evaluate the safety of administering escalating doses of banked allogeneic, partially HLA-matched rapid EBV specific T cells.
Time Frame: 8 weeks
Population: All DLT evaluable participants were included in the analysis. DLT evaluable refers to participants who received two infusions and either completed the 8 weeks toxicity evaluation period without experiencing a DLT or developed a DLT during this period. Ten participants were not evaluable for DLT and were excluded from the analysis, including one participant who was later re-enrolled and became evaluable for DLT at the 2nd enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A Cohort 1 | Group A Cohort 2 | Group A Cohort 3 | Group B Cohort 1 | Group B Cohort 2 | Group B Cohort 3 | Group C Cohort 1 | Group C Cohort 2 | Group C Cohort 3
Number analyzed (Participants) | 2 | 3 | 4 | 4 | 2 | 4 | 2 | 2 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Percent of Patients Whose Best Response is Either Complete Remission or Partial Remission
Description: To measure anti-tumor and anti-viral effects of ESTs
Time Frame: 8 weeks
Population: All response evaluable participants were included in the analysis. Participants who received the first infusion were evaluable for response, except those who received chemotherapy between the first and second infusions. Two participants were not evaluable for response and were excluded from the analysis. The participant who enrolled twice was counted as 2 individuals but was only evaluable for response at the 2nd enrollment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A Cohort 1 | Group A Cohort 2 | Group A Cohort 3 | Group B Cohort 1 | Group B Cohort 2 | Group B Cohort 3 | Group C Cohort 1 | Group C Cohort 2 | Group C Cohort 3
Number analyzed (Participants) | 2 | 3 | 6 | 5 | 3 | 7 | 2 | 3 | 3
percentage of participants | 0.0 [0.0 to 84.2] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 45.9] | 60.0 [14.7 to 94.7] | 33.3 [0.8 to 90.6] | 28.6 [3.7 to 71.0] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for 6 weeks, whereas serious adverse events were recorded for 1 year after the last EBV specific T cell infusion. All-cause mortality data were collected over a 5-year period.
Description: Adverse events were collected as per protocol for participants who received EBV Specific T cell (EST) infusions.
Arm/Group | Group A Cohort 1 | Group A Cohort 2 | Group A Cohort 3 | Group B Cohort 1 | Group B Cohort 2 | Group B Cohort 3 | Group C Cohort 1 | Group C Cohort 2 | Group C Cohort 3
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3 | 4/6 | 3/5 | 2/3 | 4/7 | 1/2 | 2/4 | 2/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 5/6 | 3/5 | 2/3 | 3/7 | 0/2 | 2/4 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 5/5 | 3/3 | 7/7 | 2/2 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A Cohort 1 (N=3) | Group A Cohort 2 (N=3) | Group A Cohort 3 (N=6) | Group B Cohort 1 (N=5) | Group B Cohort 2 (N=3) | Group B Cohort 3 (N=7) | Group C Cohort 1 (N=2) | Group C Cohort 2 (N=4) | Group C Cohort 3 (N=3)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (8) | 1 (1)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify : COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify : major hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify : Redness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify : Swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A Cohort 1 (N=3) | Group A Cohort 2 (N=3) | Group A Cohort 3 (N=6) | Group B Cohort 1 (N=5) | Group B Cohort 2 (N=3) | Group B Cohort 3 (N=7) | Group C Cohort 1 (N=2) | Group C Cohort 2 (N=4) | Group C Cohort 3 (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 4 (4) | 2 (6) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Blood and lymphatic system disorders - Other, specify : Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, specify : Clot from bleeding (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, specify : burning (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify : Hemorrhoid type bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify : sore throat (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (3) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Fever (General disorders) | 2 (3) | 1 (1) | 0 (0) | 3 (9) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify : leg cramps (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify : RSV (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify : pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify : right 2nd toe (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify : strep throat (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 4 (4) | 2 (6) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (2) | 3 (3) | 4 (6) | 3 (3) | 4 (4) | 1 (2) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 4 (12) | 1 (1) | 2 (2) | 1 (2) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 2 (2) | 2 (2) | 3 (3) | 5 (10) | 1 (1) | 3 (3) | 2 (3) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (4) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify : body aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify : dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify : tachypnea: unspecified (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify : Rash - unspecified (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify : eczematous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify : rash: unspecified (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify : unspecified rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT02287311/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT02287311/ICF_001.pdf